CLINICAL TRIAL: NCT01427101
Title: Comparison Between Cyotreductive Surgery and Debulking Surgery in Patients With Pseudomyxoma Peritonei
Brief Title: Results of CRS and Debulking in PMP Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2007/073-PMP-Andréasson
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Pseudomyxoma Peritonei
Keywords: Pseudomyxoma Peritonei; Cytoreductive surgery; Debulking surgery; Intraperitoneal chemotherapy
MeSH Terms: conditions — Pseudomyxoma Peritonei

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Patients treated from 1993 are included and during these years treatment strategy has changed. The different strategies are compared but its juts one cohort of patients. No completion date are set due to that reports from other centres show that there are longtime survivers in both treatment groups.
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to compare debulking surgery and cytoreductive surgery in patients with Pseudomyxoma Peritonei with respect to efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiology histopathology finding of Pseudomyxoma Peritonei

Exclusion Criteria:

* Preformance status WHO >2 and histopathology shows other origin then Pseudomyxoma Peritonei

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Pseudomyxoma Peritonei, sceduled for surgical treatment at Uppsala University Hospital.
Sampling Method: Probability Sample
Dates: Start 1993-09

PRIMARY OUTCOMES:
Overall survival
  from treatment and forward

SECONDARY OUTCOMES:
morbidity and mortality | 90 days
  mortality is messured during the first 90 postoperative days and morbidity during hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Haile Mahteme, MD, PhD, Principal Investigator — Uppsala University